CLINICAL TRIAL: NCT01780363
Title: MEVALONATE KINASE GENE MUTATIONS AND THEIR CLINICAL CORRELATIONS IN BEHÇET'S DISEASE
Status: Completed | Type: Observational
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Didem Arslan Tas, MD, Cukurova University
Other Study IDs: BH-MVK; CUTFBAP25011138 (Other: CUTF); CUTFBAP2501201138 (Other: CUTFBAP)
Record Dates: First submitted 2013-01-29; First posted 2013-01-31 (Estimated); Last update posted 2013-01-31 (Estimated); Status verified 2011-01

CONDITIONS: Behçet's Disease
MeSH Terms: conditions — Behcet Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- controls: frequency of mevalonate kinase gene frequency
- Behçet patients: frequency of mevalonate kinase gene mutations

SUMMARY:
Background: Genetics is suggested to play a critical role in the development of Behçet's disease (BD). Shared phenotypic features requires an approach to the differential diagnosis from periodic febrile syndromes particularly from mevalonate kinase deficiency related diseases. We planned to study for evaluating the frequency of mutations and their clinical significance in mevalonate kinase gene in Turkish patients with Behçet's disease.

ELIGIBILITY:
Inclusion Criteria:

* Behçet patients

Exclusion Criteria:

* Diagnosis of periodic fever syndromes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Turkish kindred
Sampling Method: Non-Probability Sample
Dates: Start 2011-01; Primary Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Frequency of mevalonate kinase frequency in Behçet disease | One year

SECONDARY OUTCOMES:
Mevalonate kinase gene and clinical correlations in Behçet's disease | One year

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Cukurova University, Adana
  - Didem Arslan Tas, Adana